CLINICAL TRIAL: NCT05825885
Title: The Impact of Estrogen Administration Duration on Live Birth Rates in Hormonally Prepared Frozen Embryo Transfer Cycles: a Prospective Controlled Study
Brief Title: The Impact of Estrogen Administration Duration in Hormonally Prepared Frozen Embryo Transfer Cycles
Status: Completed | Type: Observational
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, ŞAFAK OLGAN, Associate Professor, Akdeniz University
Other Study IDs: 498496942
Record Dates: First submitted 2023-04-11; First posted 2023-04-24 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Duration of Estrogen Administration
Keywords: Endometrial compaction; Endometrial receptivity; Endometrial thickness; Frozen embryo transfer; HRT; Pregnancy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- 5-7 days E2 therapy: Patient group treated with e2 for 5-7 days
- 8-10 days E2 therapy: Patient group treated with e2 for 5-7 days
- 11-13 days E2 therapy: Patient group treated with e2 for 5-7 days

INTERVENTIONS:
Drug: E2 — micronized E2 at a daily dose of 4-6mg,

SUMMARY:
This prospective controlled study aimed to investigate the effect of the duration of estrogen (E2) administration prior to progesterone (P) initiation on live birth rates (LBR) in frozen embryo transfer (FET) cycles.

The study was conducted at a single tertiary-care in vitro fertilization (IVF) center and included 486 patients undergoing high-quality frozen blastocyst transfer in a hormone replacement therapy (HRT) cycle. Patients scheduled for E2 therapy were administered either 5-7, 8-10, or 11-13 days of treatment, depending on their presentation day. After the E2-only phase, if the endometrial thickness was above 7mm, P was initiated (daily 300mg of vaginal micronized P tablets), and FET was performed on the 6th day of P treatment. The primary outcome measure was LBR.

DETAILED DESCRIPTION:
The timing of P initiation in HRT cycles depends on the thickness and morphology of the endometrium, which are influenced by the duration of E2 treatment. Although numerous studies have examined the effect of E2 treatment duration on endometrial thickness and morphology, the results have been inconsistent, and the impact on live birth rates (LBR) remains unclear. Previous research has explored the impact of standard 12-day E2 therapy and prolonged periods of E2 administration on pregnancy outcomes. However, the present study aims to compare the effects of standard 12-day E2 therapy with shorter-term E2 application and evaluate their impact on treatment outcomes.

To test hypothesis, investigators conducted a prospective analysis of about 500 hormonally prepared frozen embryo transfer (FET) cycles performed between January 2020 and December 2021 at IVF center in Akdeniz University. The objective of this study was to determine the optimal duration of estrogen (E2) therapy prior to progesterone (P) initiation for FET cycles in terms of live birth rate (LBR).

In IVF center, patients with frozen embryos routinely applied to the center on weekdays (Monday, Wednesday, and Friday) as part of a predetermined treatment plan. Patients who presented to the clinic during their menstrual periods were scheduled to receive E2 therapy for a duration of either 5-7, 8-10, or 11-13 days, depending on the day they presented. After the application of micronized E2 at a daily dose of 4-6mg, transvaginal ultrasonography was performed to assess endometrial thickness. If the endometrial thickness was found to be above 7mm, daily 300mg of vaginal micronized P tablets were initiated, and FET was performed on the 6th day of P treatment. Patients whose endometrial thickness was less than 7 millimeters on transvaginal ultrasonography after the application of E2 treatment for the specified day and who had to continue estrogen therapy were not included in the study.

The duration of E2 administration prior to P initiation was categorized into three groups: 5-7 days, 8-10 days, and 11-13 days. The primary outcome of this study was LBR, which was defined as the delivery of a live-born infant after 24 weeks of gestation. Secondary outcomes included implantation rate, clinical pregnancy rate, and miscarriage rate.

ELIGIBILITY:
Inclusion Criteria:

* Exogenous hormone preparation of the endometrial lining
* High embryo quality ((≥2BB) according to Alpha criteria
* Embryo transfer at the blastocyst stage

Exclusion Criteria:

* - Patients whose treatments were canceled for any reason before the embryo transfer procedure
* Patients who underwent embryo transfer in the cleavage stage
* Presence of low-quality (<2BB) blastocysts
* >15% loss of viability of the embryo during embryo thawing,

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: All patients who have artificial endometrial preparation with high-quality blastocysts between January 2020 and December 2021 were included.
Sampling Method: Probability Sample
Enrollment: 420 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
live birth rate | 2 years
  the birth ratio of a baby who showed any sign of life

SECONDARY OUTCOMES:
implantation rate | 2 years
  the percentage of embryos which successfully undergo implantation compared to the number of embryos transferred in a given period.
clinical pregnancy rate | 2 years
  the number of clinical pregnancy divided by the number of embryo transfer cycle for each group
miscarriage rate | 2 years
  rate of the spontaneous loss of a pregnancy before the 20th week

CONTACTS AND LOCATIONS:
Locations (1):
- Akdeniz University, Antalya, Antalya, Turkey (Türkiye)